CLINICAL TRIAL: NCT00999219
Title: FK199B (Zolpidem MR Tablet) Phase III Clinical Study - A Double-Blind, Crossover, Comparative Polysomnographic Study Using Zolpidem (Myslee®) as a Positive Control in Patients With Insomnia, Excluding Patients With Schizophrenia or Manic-Depressive Psychosis
Brief Title: A Study of FK199B to Compare Efficacy With Zolpidem by Polysomnography in Patients With Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6199-CL-0006
Record Dates: First submitted 2009-10-13; First posted 2009-10-21 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: FK199B; Zolpidem
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FK199B-first group (Experimental)
  Interventions: Drug: FK199B; Drug: Zolpidem
- Zolpidem-first group (Experimental)
  Interventions: Drug: FK199B; Drug: Zolpidem

INTERVENTIONS:
Drug: FK199B — oral
  Other Names: Zolpidem MR Tablet
Drug: Zolpidem — oral
  Other Names: Myslee

SUMMARY:
This study is to investigate the efficacy and safety of FK199B (Zolpidem MR Tablet) by polysomnography in patients with insomnia, excluding patients with schizophrenia or manic-depressive psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed as a primary insomnia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* Patients complaining of insomnia continuously for 4 weeks or longer
* Patient's usual bedtime is between 9 p.m. and 12 a.m. for the 4 week period prior to initial screening
* Patient on most occasions sleeps for a total of ≥3 and <6.5 hours over the 4 week period prior to initial screening
* Patient's usual wake time after sleep onset in a single night is ≥45 minutes per night for the 4 week period prior to initial screening
* Patients have a body weight of ≥45 kg and ≤85 kg, a BMI of ≥18.5 and <30

Exclusion Criteria:

* Patients with schizophrenia or manic-depressive psychosis
* Patients with insomnia caused by physical diseases including chronic obstructive pulmonary disease, bronchial asthma, fibrositis syndrome, chronic fatigue syndrome, rheumatic disease, climacteric disturbance, and dermatitis atopic
* Patients with circadian rhythm sleep disorder
* Patient works night shifts
* Patients with alcoholic sleep disorder
* Patients with alcohol or drug dependence or a history of these
* Patients with insomnia related with drugs including antiparkinson, antihypertensive, or steroid drugs
* Patients with sleep apnea syndrome
* Patients with restless legs syndrome or periodic limb movement disorder
* Patients with epileptic insomnia
* Patients smoke on average 40 or more cigarettes a day
* Patients who had received psychotropic drugs other than hypnotics (including anxiolytic or antidepressant drugs for hypnotic effect) within a 4 week period prior to the initial screening

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Sleep parameters estimated from polysomnography recording (wake time after sleep onset and number of awakenings) | 8 hours

SECONDARY OUTCOMES:
Mean sleep parameters estimated from polysomnography recording | 8 hours
Sleep parameters estimated from sleep questionnaire | After each night of sleep during the study period
Patient impression from sleep questionnaire | After each night of sleep during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Shikoku
  - Tōhoku